CLINICAL TRIAL: NCT01267097
Title: The PAC Study: Parents as Agents of Change in Pediatric Weight Management
Acronym: PAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: AHS Cancer Control Alberta (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Geoff Ball, Associate Professor, Department of Pediatrics, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PCWH01-2009; CIHR-MSH83715 (Other Grant/Funding Number: Funded by the Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2010-12-16; First posted 2010-12-24 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Obesity; Child
Keywords: Pediatric Obesity; Treatment; Cognitive Behavioural Therapy; Psychoeducation; Canada
MeSH Terms: conditions — Obesity; Pediatric Obesity | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioural Therapy (CBT) (Experimental): Group-based lifestyle counseling for parents
  Interventions: Behavioral: Cognitive Behavioural Therapy (CBT); Behavioral: Psycho-Education Program (PEP)
- Psycho-Education Program (PEP) (Experimental): Group-based lifestyle counseling for parents
  Interventions: Behavioral: Cognitive Behavioural Therapy (CBT); Behavioral: Psycho-Education Program (PEP)

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy (CBT) — Clinical research supports the use of CBT-based interventions in weight management for adults and children. However, the current study will advance the existing knowledge-base by combining CBT with the parents as agents of change approach for pediatric weight management. CBT is a theoretically-based therapy that focuses on the role that cognitive processes play in the maintenance of problem behaviours, mood states, and habits. CBT highlights the relationship between thoughts, feelings and actions, and utilizes techniques involving motivation, goal-setting, problem-solving, and knowledge/skill acquisition that can facilitate sustainable behaviour changes.
  Other Names: CBT
Behavioral: Psycho-Education Program (PEP) — PEP is a knowledge-based intervention that is modelled after traditional nutrition and health education programs. Research has demonstrated that knowledge based programs can improve health behaviours and outcomes in overweight and obese populations. In relation to CBT, PEP is a more passive intervention and there is limited focus on active skill building. While PEP does not represent a true control group, its content and delivery are consistent with what many clinicians provide for weight management.
  Other Names: PEP

SUMMARY:
The Canadian pediatric obesity epidemic has led to great interest in evaluating weight management care for obese children and families. Investigation is warranted since obesity is linked to risk factors for chronic diseases including type 2 diabetes mellitus (T2DM) and cardiovascular disease (CVD). Over the past 25 years, many interventions have studied the role of healthy lifestyle behaviours to help obese children achieve and maintain a healthy weight. A contemporary view of pediatric weight management interventions includes parents as a fundamental recipient of treatment. These interventions recognize the influence parents have on the lifestyle behaviours of their children. While such parent-based interventions have helped establish the role of education and behavioural theory in facilitating lifestyle changes, we believe an equally important intervention element is a focus on the role of cognitions in helping to interpret behaviour change and change maintenance. Our study incorporates cognitive behaviour theory (CBT) into an intervention for parents of obese children and compares it to a more traditional modality based on psycho-education (PEP).

Hypothesis: Obese 8 - 12 year old children (n=45) whose parents complete a 16-session, group-based, CBT intervention will achieve greater reductions in adiposity as well as improvements in physiological risk factors for T2D, lifestyle behaviours, and psychosocial outcomes at post-intervention as well as 6- and 12-months follow-up versus children (n=45) whose parents complete a 16-session, group-based, psycho-education intervention .

Primary Objective: To compare the impact of two weight management interventions (CBT versus PEP) for parents of obese children on child BMI z-score.

Secondary Objective: To measure a comprehensive set of physiological, behavioural and psychosocial outcomes in obese children and parents pre- and post-intervention.

We expect obese children whose parents complete the CBT intervention will experience greater reductions in BMI z-score vs. children whose parents complete the PEP intervention. We anticipate that improvements in parenting style, family stress, and lifestyle behaviours will be important to improve adiposity, lifestyle behaviours, and risk factors for T2DM and CVD in obese children.

ELIGIBILITY:
Inclusion Criteria: Boys and girls (n = 90) between 8 - 12 years of age with a sex- and age-specific BMI ≥95th percentile are eligible for this study. Children are referred to the Pediatric Centre for Weight and Health (PCWH) at the Stollery Children's Hospital (SCH) (Edmonton, AB, Canada) only if their BMI percentile meets or exceeds this threshold. At least one parent/guardian per family is required to participate in one of the two group-based interventions as agents of change for their family.

Exclusion Criteria: Obese children referred to the PCWH <8 years old will be referred to an outpatient dietitian for nutrition counselling; obese boys and girls >12 years old will be eligible for other weight management interventions at the PCWH. Children who do not have a parent/guardian interested in participating or possess an age- and sex-specific BMI <95th percentile will be ineligible. Children diagnosed with an endocrine disorder (i.e., Polycystic Ovarian Syndrome, Prader-Willi Syndrome, hypothyroidism) will be referred to the Endocrine Clinic at the SCH. Parents or children who are identified at screening as having severe mental health conditions or psychosocial circumstances that could limit their ability to participate in the interventions will be referred to appropriate agencies and services. Impaired ability to participate in either intervention may include substantial difficulties in attendance or implementing changes at home. Referral services may include psychological/psychiatric services, welfare services, and private nutrition or exercise counselling. Dr. Rachel Keaschuk (PCWH Psychologist and Co-I) will perform psychological interviews (75 - 90 minutes) with all families to determine family appropriateness and will lead family discussions regarding referral services (if indicated).

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2010-09; Primary Completion 2013-09 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Child BMI Z-score | Pre-intervention
Child BMI Z-score | post-intervention
Child BMI Z-score | 6-months post-intervention
Child BMI Z-score | 12-months post-intervention

SECONDARY OUTCOMES:
Lifestyle behaviours | Pre-intervention
  Nutrition (4-day food records; child and parent) and physical activity (7-day pedometer logs; child and parent) behaviours
Parental stress | Pre-intervention
  Parental stress index (PSI)
Cardiometabolic risk factors | Pre-intervention
  Blood pressure, fasting glucose, fasting insulin, HDL-C, LDL-C, total cholesterol, triglycerides (child only)
Family functioning | Pre-intervention
  Family Adaptability and Cohesion Scale-IV (FACES-IV); completed by parents
Lifestyle behaviours | post-intervention
  Nutrition (4-day food records; child and parent) and physical activity (7-day pedometer logs; child and parent) behaviours
Lifestyle behaviours | 6-months post-intervention
  Nutrition (4-day food records; child and parent) and physical activity (7-day pedometer logs; child and parent) behaviours
Lifestyle behaviours | 12-months post-intervention
  Nutrition (4-day food records; child and parent) and physical activity (7-day pedometer logs; child and parent) behaviours
Parental stress | post-intervention
  Parental stress index (PSI)
Parental stress | 6-months post-intervention
  Parental stress index (PSI)
Parental stress | 12-months post-intervention
  Parental stress index (PSI)
Cardiometabolic risk factors | post-intervention
  Blood pressure, fasting glucose, fasting insulin, HDL-C, LDL-C, total cholesterol, triglycerides (child only)
Cardiometabolic risk factors | 6-months post-intervention
  Blood pressure, fasting glucose, fasting insulin, HDL-C, LDL-C, total cholesterol, triglycerides (child only)
Cardiometabolic risk factors | 12-months post-intervention
  Blood pressure, fasting glucose, fasting insulin, HDL-C, LDL-C, total cholesterol, triglycerides (child only)
Family functioning | post-intervention
  Family Adaptability and Cohesion Scale-IV (FACES-IV); completed by parents
Family functioning | 6-months post-intervention
  Family Adaptability and Cohesion Scale-IV (FACES-IV); completed by parents
Family functioning | 12-months post-intervention
  Family Adaptability and Cohesion Scale-IV (FACES-IV); completed by parents

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Ball, PhD, RD, Principal Investigator — University of Alberta; Amanda Newton, PhD, RN, Principal Investigator — University of Alberta
Locations (1):
- Pediatric Centre for Weight and Health, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Ball GD, Mushquash AR, Keaschuk RA, Ambler KA, Newton AS. Using Intervention Mapping to develop the Parents as Agents of Change (PAC(c)) intervention for managing pediatric obesity. BMC Res Notes. 2017 Jan 13;10(1):43. doi: 10.1186/s13104-016-2361-3. PMID 28086848
- [Derived] Ball GD, Ambler KA, Keaschuk RA, Rosychuk RJ, Holt NL, Spence JC, Jetha MM, Sharma AM, Newton AS. Parents as agents of change (PAC) in pediatric weight management: the protocol for the PAC randomized clinical trial. BMC Pediatr. 2012 Aug 6;12:114. doi: 10.1186/1471-2431-12-114. PMID 22866998
- See also: Pediatric Centre for Weight and Health — http://www.albertahealthservices.ca/services.asp?pid=service&rid=1004154